CLINICAL TRIAL: NCT03774498
Title: Effect of Different Over-the-counter Toothpastes on Enamel Remineralization: A Double Blinded Randomized Clinical Trial
Brief Title: Effect of Different Over-the-counter Toothpastes on Enamel Remineralization
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Farag Abd El-Khalek kelany, Principal investigator, Cairo University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-11-22
Record Dates: First submitted 2018-12-10; First posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Enamel Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensodyne repair and protect (Active Comparator): NovaMin & fluoride toothpaste
  Interventions: Drug: Sensodyne repair and protect
- Sensodyne Daily Care Toothpaste 0.315% (No Intervention): Sodium fluoride toothpaste

INTERVENTIONS:
Drug: Sensodyne repair and protect — NovaMin & fluoride toothpaste
  Other Names: no other names
  Arms: Sensodyne repair and protect

SUMMARY:
This study will be conducted to compare between recent over-the-counter toothpaste (Novamin & Fluoride) and regular over-the-counter toothpaste (Sodium Fluoride) in remineralization potential, so as to be able to know which of the toothpastes will have a better remineralization potential on demineralized enamel.

DETAILED DESCRIPTION:
Statement of problem:

Dental caries has been recognized as a dynamic process that results from an imbalance between the physiologic demineralization and remineralization of tooth structure. It has been well established that tooth undergoes cyclic demineralization of enamel crystals with periods of remineralization resulting from re-precipitation of calcium and phosphate ions from the saliva. If the process of demineralization dominates, caries result. However, if remineralization dominates along with removal of bacterial infection, enamel integrity gets restored. This basic knowledge of carious process brings us to an understanding that by controlling the amount, pattern and rhythm of demineralization and remineralization, carious lesions can either be controlled from progressing further or can be reversed. Several decades ago it was noted that clinically detectable white-spot lesions could be hardened; various scientific methods have been advocated for arrest and the reversal of incipient caries lesion by either decreasing the solubility of the mineral present or by increasing the mineral content of the previously demineralized tooth. Since remineralization occurring naturally in oral environment is often inadequate for maintaining strong decay free enamel and dentin, the process needs to be augmented by using some external means. It has been proposed that a simultaneous supply of calcium, phosphate and fluoride ions might serve as an invaluable tool to remineralize and strengthen the tooth structure by formation of calcium fluorapatite. Fluoride as a constituent of drinking water and in the form of various topically applied products especially over-the-counter toothpastes have a long successful history of use as a caries preventive agent.

NovaMin is claimed to release calcium and phosphate ions intraorally to help the self-repair process of enamel. A silica-rich surface layer forms through poly-condensation of hydrated silica groups on which precipitation of ions happens which crystallizes over time to form a hydroxyl-carbonate apatite. Although it is used extensively as a desensitizing agent reports also claim that the chemical reactions that promote apatite formation may enhance the remineralization. But there is limited clinical research to ascertain if there is any synergistic effect on combining anti-cariogenic activity of fluoride ions with these remineralization systems.

Direct benefit of the research to the human volunteer:

* Have better remineralization for initial white spot carious lesions using recent Novamin technology.
* Gain the other advantages for Novamin technology on the gingival health as well as dental health.
* Patient will know the proper brushing technique as he would be given instructions about this during the study.
* Patient will get to know the difference in efficiency of different over-the-counter toothpastes especially those assigned in the investigator's study.

Scientific value and social Benefits:

* Determine whether the new Novamin technology results are worth and have good efficient remineralization potential or not.
* Know more conservative mean for repair of demineralized areas in teeth.
* Have proper data base about difference in over-the-counter toothpastes.

Research question:

Will recent over-the-counter toothpaste (Novamin & Fluoride) be better than regular over-the-counter toothpaste (Sodium Fluoride) in remineralization of white spot lesions in adult patients who are having initial white spot carious lesions?

ELIGIBILITY:
Inclusion Criteria:

* Patients having at least two permanent tooth surfaces having white spot lesions (buccal/facial aspects of incisors, canines or pre-molars).
* Subjects with orthodontic appliances.
* Systemically healthy subjects of both genders, between the ages of 18 to 45 years, who were well versed with the use of toothbrush and dentifrice for oral hygiene maintenance, will be considered for the study.

Exclusion Criteria:

* Presently on desensitizing treatment.
* Subjects with bridge work that may interfere with evaluation.
* Medical histories that may compromise study protocol.(including psychiatric and pharmaco-therapeutic problems)
* Allergies.
* Systemic conditions which are etiologic/predisposing to dentinal hypersensitivity (Enamel and dentine genetic abnormalities).
* Eating disorders.
* Pregnancy or breast feeding.
* Any other pathology.
* Known history of allergies to toothpaste contents.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Enamel remineralization | 8 weeks
  Decalcification index: (0):No white spot ,(1):Visible white spots ,no surface interruption (mild),(2):Visible white spot with roughened surface,not require restoration (moderate),(3):Visible with surface interruption (severe), (4):Cavitation.
  International Caries Detection and Assessment System:(0):Sound tooth surface: No evidence of caries after 5 sec air drying ,(1):First visual change in enamel: Opacity or white or brown discoloration visible after prolonged drying,(2):Distinct change in enamel visible when wet, must be visible when dry,(3):Localized enamel breakdown (no visual signs of dentin involvement) seen when wet and after prolonged drying,(4):Underlying dark shadow from dentine,(5):Distinct cavity with visible dentine,(6): Extensive (more than half the surface) cavity with visible dentine.
  Scoring is done by photographs at the beginning and at follow-up visits with the same setting each time.

CONTACTS AND LOCATIONS:
Overall Officials: Omyma Safwat, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided